CLINICAL TRIAL: NCT04674085
Title: Real-life Experience of Tofacitinib in Patients With Treatment-Resistant Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sibel Ocak Serin, Principal Investigator, Umraniye Education and Research Hospital
Other Study IDs: Umraniye ERH
Record Dates: First submitted 2020-12-06; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Rheumatoid Arthritis; Treatment Adherence and Compliance
Keywords: Rheumatoid Arthritis; tofacitinib; disease activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to present the efficacy and safety data for patients with RA who received tofacitinib therapy in outpatient clinics.

DETAILED DESCRIPTION:
This retrospective cohort study included 35 patients with rheumatoid arthritis who received tofacitinib therapy in rheumatology outpatient clinic between June 2015 and December 2019. Patients who received tofacitinib due to unresponsiveness to ≥2 conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) and/or ≥1 biological disease-modifying anti-rheumatic drugs (bDMARDs) were retrospectively evaluated. Demographic characteristics of the patients, the disease activity score-28 for rheumatoid arthritis with erythrocyte sedimentation rate (DAS 28-4 (ESR)), change in DAS-28, health assessment questionnaire score, visual analogue scale score, and laboratory parameters such as erythrocyte sedimentation rate (ESR), C-reactive protein (CRP) level, hemogram, lipid parameters, and uric acid were recorded. The data at six months of treatment were compared with baseline data. The effects related to the treatment as well as the undesired consequences were evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients who received tofacitinib due to unresponsiveness to ≥2 csDMARDs and/or ≥1 bDMARDs were retrospectively evaluated.

-

Exclusion Criteria:

Patients who could not tolerate the treatment and whose follow-up results could not be reached were excluded from the study.

-

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort study
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluates the effects of tofacitinib therapy by measuring change in DAS 28-4 (ESR) and improvement in DAS-28 | 6 months
  Clinical and laboratory parameters (DAS 28-4 (ESR), improvement in DAS-28) will be compared at the end of six months with baseline data in patients with rheumatoid arthritis refractory to conventional synthetic disease-modifying anti-rheumatic drugs and/or biological disease-modifying anti- rheumatic drugs.
Evaluates the effects of tofacitinib therapy by measuring change in health assessment questionnaire score, visual analogue scale score | 6 months
  Clinical parameters (health assessment questionnaire score, visual analogue scale score) will be compared at the end of six months with baseline data in patients with rheumatoid arthritis refractory to conventional synthetic disease-modifying anti-rheumatic drugs and/or biological disease-modifying anti- rheumatic drugs.
Evaluates the effects of tofacitinib therapy by measuring change in erythrocyte sedimentation rate (ESR) | 6 months
  Laboratory parameters (erythrocyte sedimentation rate (ESR)) will be compared at the end of six months with baseline data in patients with rheumatoid arthritis refractory to conventional synthetic disease-modifying anti-rheumatic drugs and/or biological disease-modifying anti- rheumatic drugs.
Evaluates the effects of tofacitinib therapy by measuring change C-reactive protein (CRP) level | 6 months
  Laboratory parameters (C-reactive protein (CRP) level) will be compared at the end of six months with baseline data in patients with rheumatoid arthritis refractory to conventional synthetic disease-modifying anti-rheumatic drugs and/or biological disease-modifying anti- rheumatic drugs.
Evaluates the effects of tofacitinib therapy by measuring change hemogram | 6 months
  Laboratory parameters (hemogram) will be compared at the end of six months with baseline data in patients with rheumatoid arthritis refractory to conventional synthetic disease-modifying anti-rheumatic drugs and/or biological disease-modifying anti- rheumatic drugs.
Evaluates the effects of tofacitinib therapy by measuring change lipid parameters | 6 months
  Laboratory parameters (lipid parameters , Total Cholesterol; LDL, Low-Density Lipoprotein; HDL, High-Density Lipoprotein; TG, triglyceride) will be compared at the end of six months with baseline data in patients with rheumatoid arthritis refractory to conventional synthetic disease-modifying anti-rheumatic drugs and/or biological disease-modifying anti- rheumatic drugs.
Evaluates the effects of tofacitinib therapy by measuring change uric asid | 6 months
  Laboratory parameters (uric asid) will be compared at the end of six months with baseline data in patients with rheumatoid arthritis refractory to conventional synthetic disease-modifying anti-rheumatic drugs and/or biological disease-modifying anti- rheumatic drugs.